CLINICAL TRIAL: NCT00282321
Title: High-protein and High-carbohydrate Diets' Effect on Urinary Concentrating Ability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2006.01.TGK
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — Diet, High-Protein; Diet, High-Protein Low-Carbohydrate

INTERVENTIONS:
Behavioral: High Protein diet
Behavioral: High carbohydrate diet

SUMMARY:
We wanted to test urinary concentrating ability and AQP-2 expression in kidney during high-protein and high-carbohydrate diet.

ELIGIBILITY:
Inclusion Criteria:

* (1) Genders; both mal and female
* (2) Age; 18- 65 years old
* (3) BMI; below 30
* (4) Females had to bee in oral contraceptive treatment

Exclusion Criteria:

* (1) Clinical signs or history of disease in the heart, lungs, kidneys or endocrine organs
* (2) Abnormal laboratory test (blood haemoglobin, white cell count, platelets, plasma sodium, plasma potassium, plasma creatinine, plasma albumin, plasma bilirubin, plasma alanine aminotransferase, plasma cholesterol and blood glucose)
* (3) Albuminuria or glucosuria
* (4) Cancer
* (5) Arterial hypertension
* (6) Alcohol abuse
* (7) Use of tobacco
* (8) Medical treatment, except oral contraceptives
* (9) Pregnancy or breast feeding
* (10) Medicine abuse
* (11) Donation of blood less than 1 month before the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
u-AQP-2
FeNa+

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Holstebro Hospital, 7500 Holstebro Denmark; Thomas G Knudsen, MD, Principal Investigator — Holstebro Hospital, 7500 Holstebro, Denmark
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Denmark